CLINICAL TRIAL: NCT01652144
Title: A Phase II Study of AT7519M, a CDK Inhibitor, in Patients With Relapsed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I194
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-03

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AT7519M (Experimental): AT7519M: 27 mg/m2 IV injection, 1 hour infusion, 27 mg/m2/day twice weekly x 2 weeks every 3 weeks (days 1, 4, 8 and 11)
  Interventions: Drug: AT7519M

INTERVENTIONS:
Drug: AT7519M

SUMMARY:
The purpose of this study is to find out what effects a new drug AT7519M has on mantle cell lymphoma.

DETAILED DESCRIPTION:
This research is being done because AT7519M has been shown to shrink tumours in animals and has been studied in a few people and seems promising but it is not clear if it can offer better results than standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented mantle cell lymphoma non-refractory to prior therapy. Diagnosis of mantle cell lymphoma should be confirmed by the local institution's lymphoma pathologist.
* Presence of clinically and/or radiologically documented disease. At least one site of disease must be bidimensionally measurable using CT or MRI performed in the 3 weeks prior to study enrolment. Bone lesions are not considered to be bidimensionally measurable.
* Minimum size of at least ONE lesion must be as follows: (must be done within 21 days prior to registration)
* Lymph nodes (measured by spiral CT scan) > 1.5 cm x or 1.5 cm

Other non-nodal lesions:

MRI ≥ 1 cm x 1 cm CT scan ≥ 1 cm x 1 cm Physical exam ≥ 1 cm x 1 cm (e.g. skin lesion, nodules)

* Patients must have a life expectancy of at least 12 weeks.
* Age ≥ 18 years.
* ECOG performance status of 0, 1 or 2 (see Appendix II).
* Previous Therapy Patients must have received at least one, and up to three prior systemic chemotherapy regimens (high dose chemotherapy with autologous stem cell support is permitted but this must be counted as one line of therapy) but must NOT have shown disease progression while receiving chemotherapy or within 1 month of last dose of most recent therapy (i.e. must be non-refractory).

Systemic Therapy:

Patients must be ≥ 4 weeks since last dose of systemic therapy (including investigational). As noted, 1-3 previous chemotherapy regimens may have been given. NB: The same chemotherapy combination given for first line therapy and second line therapy is considered two regimens. Exceptions to the 4-week interval since last treatment are possible if prior therapy is non-myelosuppressive or if any treatment-related myelosuppression has resolved.

Not permitted:

* Radioactive Monoclonal Antibody Therapy
* Prior treatment with AT7519M or another CDK inhibitor
* Previous allogeneic stem cell transplant (Note: autologous stem cell transplant is permitted) Prior rituximab or bortezomib treatment is permitted, but they must be counted as systemic therapy regimens if given as single agents.

Radiation:

Patients may have had radiation, provided a minimum of 21 days has elapsed prior to enrollment. Patients must have recovered from any acute toxic effects from radiation prior to registration.

Surgery:

Previous surgery is permitted provided that wound healing has occurred and at least 14 days have elapsed if surgery was major.

* Laboratory Requirements: (must be done within 7 days prior to registration) Hematology Absolute neutrophils (ANC) ≥ 1.0 x 109/L Platelets ≥ 75 x 109/L Chemistry Serum creatinine ≤ UNL Bilirubin ≤ UNL AST and ALT ≤ 2.5 x UNL Potassium, calcium, magnesium - Within normal limits Creatine Kinase (CK or CPK) ≤ UNL
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. The patient must sign the consent form prior to registration.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient registration.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 5 years.
* Patients with known CNS involvement by lymphoma. Tests to investigate CNS involvement are required only if clinically indicated (i.e. disease suspected on basis of symptoms or other findings).
* Patients with known hypersensitivity to the study drug or its components.
* The following are exclusions for enrolment on the study:

  1. Pregnant or lactating women. (N.B.: All women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to registration).
  2. Men and women of childbearing potential who do not agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of the study participation. (Should a woman become pregnant or suspect she is pregnant, or should a man father a child, while participating in this study, she/he should inform the treating physician immediately.)
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including, but not limited to:

  1. history of significant neurologic or psychiatric disorder (e.g. uncontrolled psychotic disorders) which would impair the ability to obtain consent or limit compliance with study requirements;
  2. active uncontrolled or serious infection;
  3. pulmonary disease requiring oxygen;
  4. known HIV infection or other immune deficiency;
  5. other medical conditions that might be aggravated by study treatment
* Patients with pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction as follows:

  1. Significant cardiac event (including symptomatic heart failure or angina) within 3 months of entry or any cardiac disease that, in the opinion of the investigator, increases risk for ventricular arrhythmia.
  2. Any personal history of ventricular arrhythmia, which was symptomatic or required treatment (CTC grade 3). This includes: multifocal PVCs, bigeminy, trigeminy, ventricular tachycardia)
  3. Uncontrolled hypertension (systolic blood pressure of 150 mmHg or higher or diastolic blood pressure of 95 mmHg or higher)
  4. A previous history of drug induced significant QTc prolongation (defined as a QTc interval equal to or greater than 500msec) or causing significant ECG abnormalities
  5. Congenital long QT syndrome
  6. QT and QTc, unmeasurable or > 460 msec on screening ECG
  7. Left ventricular ejection fraction of less than the institution's lower limit of normal (LLN) measured by MUGA or echocardiogram
* Patients who are currently receiving treatment with agents with a known risk of Torsades de Pointes. (see http://torsades.org (list #1)). However, patients may be enrolled on study if treatment with such agents is stopped ≥ 7 days prior to first dose of AT7519M.
* Patients with pre-existing peripheral neuropathy (sensory and/or pain) > grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09-14 (Actual); Primary Completion 2014-12-02 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Efficacy | 24 months
  objective response rate of AT7519M when given as a 1 hour intravenous infusion twice weekly for two out of three weeks in patients with relapsed mantle cell lymphoma (MCL).

SECONDARY OUTCOMES:
Severity of toxicity | 24 months
Time to progression | 24 months
Response duration | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: John Kuruvilla, Study Chair — Univ. Health Network-Princess Margaret Hospital
Locations (6):
- Canada (6):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seftel MD, Kuruvilla J, Kouroukis T, Banerji V, Fraser G, Crump M, Kumar R, Chalchal HI, Salim M, Laister RC, Crocker S, Gibson SB, Toguchi M, Lyons JF, Xu H, Powers J, Sederias J, Seymour L, Hay AE. The CDK inhibitor AT7519M in patients with relapsed or refractory chronic lymphocytic leukemia (CLL) and mantle cell lymphoma. A Phase II study of the Canadian Cancer Trials Group. Leuk Lymphoma. 2017 Jun;58(6):1358-1365. doi: 10.1080/10428194.2016.1239259. Epub 2016 Oct 17. PMID 27750483